CLINICAL TRIAL: NCT06175962
Title: The Effect of The Menopause Adaptatıon Program Developed Based on Meleıs' Transıtıon Theory, on The Attıtudes Towards Menopause And Spırıtual Well-Beıng of Perımenopusal Women
Brief Title: Perımenopausal Women's Attıtudes Towards Menopause and Spırıtual Well-Beıng
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sinop University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SINOPUakufaci
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Menopause; Activity, Motor; Attitude
Keywords: Perimenopause; Baduanjin; Menopause attitude
MeSH Terms: conditions — Motor Activity; Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): At the beginning of the research, the Introductory Information Form, the Attitudes Towards Menopause Scale (MITÖ), and the Spirituality Index Well-Being Scale will be applied to the experimental group. Later, menopause health education will be given to women within the scope of the menopause adaptation program prepared based on Meleis's transition theory. Then, the women will be taught the baduanjin exercise for 4 weeks by the researcher who has a Qigong practitioner certificate. All training will be held online. After making sure that the women have learned the baduanjin exercise, they will be asked to do the baduanjin exercises at home 3 times a week for 8 weeks.
  During this process, counseling services will be provided and women will be followed. The study will be completed in 14 weeks, after which posttest data will be collected.
  Interventions: Behavioral: TRAINING AND EXERCISE
- Control Group (No Intervention): At the beginning of the research, the Introductory Information Form, Attitudes Towards Menopause Scale (MITÖ), and Spirituality Index Scale will be applied to the control group.
  No intervention will be made to the control group.

INTERVENTIONS:
Behavioral: TRAINING AND EXERCISE — Menopause health training will take place in 2 sessions each week and will be completed in 4 sessions. Each session duration is 45 minutes. Baduanjin exercise training will take place in 2 sessions per week, each session lasting 30 minutes. It will be completed in 8 sessions in total. Relaxing music will be played during the Baduanjin exercise and relaxation will be encouraged. During the Baduanjin exercise, proper posture, conscious breathing and focus of the mind will be prioritized. While the movements are being implemented, their symbolic meanings will be explained to the participants. Women will be asked to perform baduanji 3 times a week for 8 weeks.
  During this process, reminder messages will be sent to women via WhatsApp.
  Arms: Experimental Group

SUMMARY:
Menopause; cessation of menstruation due to cessation of follicular activity is the transition from the reproductive period to non-reproductive life. Considering that the average life expectancy is increasing, women spend most of their lives in the menopausal period. Women who have a positive attitude towards menopause have a positive body image, experience less depressive experiences, and the severity of menopause symptoms decreases. It has also been assumed that spiritual well-being is effective in reducing the severity of menopause symptoms and anxiety, supporting positive body image, and coping with losses.

Baduanjin exercise is a type of body mind exercise. It increases the production of life energy and distributes it to different aspects of the body.

It is thought that the baduanjin body-mind exercise to be applied to perimenopausal women will have positive effects on the spiritual well-being of menopausal women and their attitudes towards menopause. Thus, it is expected that women's transition and adaptation to the menopause process will be easier.

DETAILED DESCRIPTION:
This study will be carried out as a pre-test - post-test randomized controlled experimental study. The population of the research consists of female patients between the ages of 45-55 who are registered to a family health center located in a provincial center in the north of Turkey. Women who are in the perimenopausal period and meet the inclusion criteria according to the Staging of Reproductive Aging in Women (STRAW) criteria will be included in the study. The random.org program will be used to unbiasedly assign 60 women who meet the research criteria to the experimental and control groups.

The menopause adaptation program will be applied to the intervention regimen. This program, which will be applied to the experimental group, was prepared based on the Meleisin Transition theory. Since women's menopause is a transition process, the transition theory was preferred. Within the scope of the program, the experimental group will be given online menopause health education for the first 6 weeks and baduanjin exercise will be taught. For the next 8 weeks, individuals will be asked to practice the baduanjin exercise 3 times a week. Online consultation will be provided during this period.

The study will be completed in 14 weeks in total. No intervention will be applied to the control group. The study will be terminated after the post-test data is collected. Data will be collected using the Introductory Information Form, the Attitudes Towards Menopause Scale (MITÖ, Spirituality Index of Well-Being Scale).

ELIGIBILITY:
Inclusion Criteria:

* Being in the perimenopausal period
* Being between the ages of 40-55
* Having entered menopause naturally
* Volunteering to participate in research

Exclusion Criteria:

* Having a physical problem that prevents exercise
* Being on hormone therapy
* Not having a menstrual period for more than 8 months
* Not using a smartphone

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women in the perimenopausal period according to the Staging of Reproductive Aging in Women (STRAW) criteria
Enrollment: 60 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Attitude Scale towards Menopause (MITÖ) | 14 WEEKS
  It was developed by Uçanok (1994) to measure the attitudes of women in different age groups towards menopause and its aftermath. There are a total of 20 statements in the scale, 2 positive and 18 negative. The scale is a four-point Likert type. For negative expressions, scoring is done in the opposite direction. The lowest score that can be obtained from the scale is 0 and the highest score is 80. It is accepted that the higher the scores above the average score of 40, the more positive the attitude.

SECONDARY OUTCOMES:
Spirituality Index of Well-Being Scale | 14 WEEKS
  Keskinoğlu et al. (2019) conducted the Turkish validity and reliability study of the scale developed by Daaleman and Frey (2004). The scale is a 5-point Likert type consisting of 2 sub-dimensions and 12 items. All items of the scale, which have sub-dimensions of self-efficacy 1, 2, 3, 4, 5, 6 (6 items) and Life schema 7, 8, 9, 10, 11, 12 (6 items), were prepared in reverse and scored in reverse. A high score from each sub-dimension of the scale shows that the individual has the characteristic evaluated by the relevant sub-dimension. The scale also gives a total well-being score. An increase in the scale score indicates an increase in spiritual well-being. When scoring the scale, the average of the sub-dimensions and the total score is taken.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur ATAMAN KUFACI, Principal Investigator — Sinop University
Locations (1):
- Aynur ATAMAN KUFACI, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No